CLINICAL TRIAL: NCT00221728
Title: Treatment of Renal Tumors With Radiofrequency: Efficacy Evaluation in Comparison With Conservative Surgery (Multicentric Randomized Trial)
Brief Title: Comparison Between Surgery and Radiofrequency for Treatment of Renal Tumors
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: lack of patients
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Ministry of Health, France (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9359-03; 2003-006
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2010-05-28 (Estimated); Status verified 2010-05

CONDITIONS: Kidney Neoplasms
Keywords: Kidney Neoplasms; Surgery; Catheter Ablation; Randomized controlled trials; Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Neoplasms; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Radiofrequency
Procedure: conservative surgery

SUMMARY:
Surgical treatment of multiple or recurrent renal tumors may be complicated by renal function impairment. Mini-invasive thermotherapy as radiofrequency (RF), induces necrosis of tumoral tissue while sparing normal renal parenchyma. The purpose of the study is to compare, in patients at risk of renal insufficiency, a strategy based on surgical approach and a strategy based on RF approach. 180 patients from 9 centers will be randomized in two groups (surgical vs. RF, delivered either percutaneously or under laparoscopy). The proportion of patients with a local carcinologic efficacy at 5 years and the general and renal tolerance will be analysed and compared between both strategies.

DETAILED DESCRIPTION:
Background. Surgical treatment of multiple or recurrent renal tumors may be complicated by renal function impairment. Mini-invasive thermotherapy as radiofrequency (RF), induces necrosis of tumoral tissue while sparing normal renal parenchyma.

Objectives. The main objective is to assess the 5-year local carcinologic efficacy (no residual tumor tissue and no recurrence at the site of treatment) of the radiofrequency treatment. Secondary objectives are to assess 5-year overall carcinologic efficacy, predictive factors of technical success of RF procedures, and the general and renal tolerance 5 years after treatment.

Study design. Open label, randomized, parallel-group, multicentric clinical trial (9 centers).

Eligibility criteria. Patients with renal tumor in whom a surgical treatment may result in renal function impairment.

Intervention.

Experimental group: radiofrequency treatment, percutaneous or under laparoscopy, using RF 3000™ generator (Radiotherapeutics, Boston scientific) under a standardized heating protocol. A second procedure is allowed in case of residual tumoral tissue or tumor recurrence.

Control group: conservative kidney surgery.

Outcomes. The principal outcome is the 5-year local carcinologic efficacy (no residual tumor tissue and no recurrence at the site of treatment, as assessed by tomodensitometry or MRI after injection). Secondary outcomes are 5-year overall carcinologic efficacy (local efficacy and no metastases), renal function, technical success of RF procedures (no residual tumor tissue 2 months after procedure) and tolerance.

Follow-up. Clinical, biological and imaging follow-ups are scheduled 2 months, 6 months, 1, 2, 3, 4 and 5 years after the first treatment.

ELIGIBILITY:
Inclusion Criteria:

* Solid kidney tumor: diameter <= 40mm, maximum volume 32cc
* Intra-parenchymatous localization
* At least one of the following criteria:

  * Patient of more than 70 years old
  * Hereditary kidney cancer (von Hippel-Lindau Disease disease, hereditary tubulopapillary carcinoma...)
  * Single kidney, with tumor difficult to reach to a conservative surgery (central-hilar or intra-parenchymatous tumour...)
  * Context of local recurrence after partial kidney surgery
  * Patient with impaired renal function (renal clearance < 30 ml/min)
* Written informed consent

Exclusion Criteria:

* Conservative surgery feasible in good technical and carcinological conditions
* Contra-indication to either treatment
* Kidney cancer metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2005-04; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Estimated)

PRIMARY OUTCOMES:
Carcinologic efficacy at the site of treatment, | at 5 years

SECONDARY OUTCOMES:
Overall carcinologic efficacy | at 5 years
Carcinologic efficacy and lack of adverse consequences on renal function | at 5 years
Local technical success

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Grenier, Professor, Principal Investigator — University Hospital, Bordeaux; Arnaud Méjean, Professor, Principal Investigator — Hôpital Necker, Paris; Paul Perez, Dr, Study Chair — University Hospital, Bordeaux
Locations (1):
- Service de radiologie B, Hôpital Pellegrin, Bordeaux, France